CLINICAL TRIAL: NCT03930173
Title: A Prospective Pilot to Evaluate the Diagnostic Assessment of 18F-Fluciclovine Positron Emission Tomography to Distinguish Tumor Progression From Radiation Necrosis Following Stereotactic Radiosurgery for Brain Metastases
Brief Title: 18F-Fluciclovine PET to Distinguish Tumor Progression From Radiation Necrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE2319
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Secondary Malignant Neoplasm of Brain and Cerebral Meninges
MeSH Terms: conditions — Brain Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 18F-fluciclovine PET/CT of the brain (Experimental): Arm includes participants with a known diagnosis of brain metastases who have undergone prior intracranial SRS and whose MRI brain scan is equivocal for radiation necrosis versus tumor progression.
  Participants will undergo 18F-fluciclovine PET/CT of the brain. Qualitative and quantitative metrics will be documented at the time of image acquisition. Qualitative image assessment will be performed independently by 3 separate physicians.
  Interventions: Drug: 18F-fluciclovine; Device: PET/CT of the brain

INTERVENTIONS:
Drug: 18F-fluciclovine — A single dose of 18F-fluciclovine will be administered intravenously for PET/CT imaging. The standard 10 mCi dose will be used for this study.
Device: PET/CT of the brain — Each subject will undergo 18F-fluciclovine PET/CT of the brain which will be performed ≤ 30 days from equivocal MRI brain

SUMMARY:
The purpose of this study is to evaluate whether 18F-fluciclovine PET/CT of the brain, is able to distinguish radiation necrosis from tumor progression in cases where MRI is inconclusive.

18F-fluciclovine is an FDA approved radioactive diagnostic agent and is injected into the participant and then taken up by cancer cells, which can then be visualized with a PET/CT scan. 18F-fluciclovine is FDA approved for the detection of recurrent prostate cancer, but is still investigational for the purposes of this study.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the accuracy of 18F-fluciclovine PET in distinguishing radiation necrosis from tumor progression. Accuracy will be assessed via receiver operating characteristic curve analysis, as well as by calculating sensitivity and specificity.

Secondary objectives of this study are to assess which factors may influence accuracy of 18Ffluciclovine PET in distinguishing radiation necrosis from tumor progression and to compare the accuracy of each of the qualitative and quantitative metrics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a confirmed diagnosis of brain metastases.
* Subjects must have received prior intracranial SRS at least once for brain metastases. Prior WBRT is allowed.
* Subjects must have had a clinical tumor protocol MRI of the brain including a DSC-MR perfusion sequence, which is equivocal for radiation necrosis versus tumor progression within 30 days of treatment scan. "Equivocal" will be defined as being inconclusive for radiation necrosis versus tumor progression as determined by the study neuroradiologist.
* Physician assessed life expectancy of ≥ 6 months.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential, a negative serum pregnancy test within 14 days of registration is required.

Exclusion Criteria:

* Subjects who have experienced a prior anaphylaxis reaction to 18Ffluciclovine are not eligible.
* Females pregnant at the expected time of 18F-fluciclovine administration are not eligible due to potential harm to the fetus from exposure to radiation. Women who could be pregnant require a negative pregnancy test to be eligible.
* Women who are breast feeding at the expected time of 18F-fluciclovine administration are not eligible due to potential harm to the infant from exposure to radiation.
* Subjects contraindicated for MRI.
* Subjects unable or unwilling to comply with study requirements are not eligible.
* Major medical illness or psychiatric impairments, which in the investigator's opinion, will prevent completion of protocol therapy and/or preclude informed consent.
* Brain metastases from primary lymphoma, germ cell tumor, or small cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of 18F-fluciclovine PET as measured by area under the ROC curve (AUC) | Up to 1 year from start of study
  The accuracy of 18F-fluciclovine PET in distinguishing radiation necrosis from tumor progression will be reported. Accuracy will be assessed via receiver operating characteristic curve analysis.

SECONDARY OUTCOMES:
18F-fluciclovine uptake in lesions, compared to normal brain tissue. | Up to 1 year from start of study
  18F-fluciclovine uptake in lesions will be reported in comparison to normal brain tissue.
Sensitivity and specificity of 18F-fluciclovine PET | Up to 1 year from start of study
  Sensitivity and specificity of 18F-fluciclovine PET diagnostic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Chao, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125